CLINICAL TRIAL: NCT03759366
Title: An Open-Label, Multicenter Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Eculizumab in Pediatric Patients With Refractory Generalized Myasthenia Gravis
Brief Title: A Phase 3 Open-Label Study of Eculizumab in Pediatric Participants With Refractory Generalized Myasthenia Gravis (gMG)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECU-MG-303; 2016-001384-37 (EudraCT Number)
Record Dates: First submitted 2018-11-26; First posted 2018-11-30 (Actual); Results first posted 2022-08-25 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Myasthenia Gravis; Myasthenia Gravis, Juvenile Form; Myasthenia Gravis, Generalized
Keywords: Myasthenia Gravis; Myasthenia Gravis, Generalized
MeSH Terms: conditions — Myasthenia Gravis | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eculizumab Intravenous (IV) Infusion (Experimental): In the Primary Evaluation Treatment Period (26 weeks), eculizumab will be administered weekly during the initial induction phase and every 2 weeks during the maintenance phase.
  In the Extension Period (up to 208 weeks), participants will continue to receive eculizumab every 2 weeks.
  Eculizumab will be administered at doses of 300, 600, 900, or 1200 milligrams (mg), based on the participant's current body weight.
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Eculizumab will be administered by IV infusion.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, pharmacokinetics, and pharmacodynamics of eculizumab in the treatment of pediatric refractory gMG based on change from Baseline in the Quantitative Myasthenia Gravis (QMG) score for disease severity.

DETAILED DESCRIPTION:
The study will consist of an up to 4-week Screening Period, 26-week Primary Evaluation Treatment Period, an additional (up to) to 208-week Extension Period, and an 8-week Safety Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female pediatric participants 6 to <18 years of age at time of assent/consent.
* Vaccinated against Neisseria meningitidis.
* Documented vaccination against Haemophilus influenzae and Streptococcus pneumoniae infections prior to dosing as per local and country specific immunization guidelines for the appropriate age group.
* Diagnosis of MG confirmed by positive serologic test for anti-acetylcholine receptor antibodies at Screening, and 1 of the following: (a) history of abnormal neuromuscular transmission test demonstrated by single-fiber electromyography or repetitive nerve stimulation; (b) history of positive anticholinesterase test (for example, edrophonium chloride or neostigmine test); or (c) participant demonstrated improvement in MG signs on oral acetylcholinesterase inhibitors, as assessed by the Investigator.
* Presence of refractory gMG, defined as participants with gMG who have 1 or more of the following: (a) failed treatment ≥1 year with at least 1 immunosuppressive therapies (IST), defined as follows: (1) persistent weakness with impairment of activities of daily living; (2) myasthenia gravis (MG) exacerbation and/or crisis while on treatment; or (3) intolerance to ISTs due to side effect or comorbid condition(s). (b) Require maintenance plasma exchange (PE) or intravenous immunoglobulin (IVIg) to control symptoms; and/or (c) in the opinion of the Investigator, MG poses a significant functional burden despite current MG treatment.
* MGFA Clinical Classification of Class II to IV at Screening.
* In patients aged 12 to 18 years, QMG total score ≥ 12 at Screening; in patients aged 6 to 11 years, no minimum QMG is required for inclusion; however, patients must have documented limb weakness in at least one limb.
* All MG-specific treatment has been administered at a stable dosing regimen of adequate duration prior to Screening.

Exclusion Criteria:

* Parent or legal guardian is an Alexion employee.
* Any active or untreated thymoma. History of thymic carcinoma or thymic malignancy unless deemed cured by adequate treatment with no evidence of recurrence for ≥5 years before Screening.
* History of thymectomy within 12 months prior to Screening.
* Are pregnant or lactating.
* Any unresolved acute, or chronic, systemic bacterial or other infection, which is clinically significant in the opinion of the Investigator and has not been treated with appropriate antibiotics.
* Use of PE within 4 weeks prior to first dose.
* Use of rituximab within 6 months prior to first dose.
* Patients who are under 15 kg and are receiving maintenance IVIg.
* Participation in another interventional treatment study or use of any experimental therapy within 30 days before initiation of study drug on Day 1 in this study or within 5 half-lives of that investigational product, whichever is greater.
* Have previously received treatment with eculizumab or other complement inhibitors.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2023-11-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (8):
  - Research Site, Los Angeles, California
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Columbia, Missouri
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
- Japan (3):
  - Research Site, Iruma-Gun
  - Research Site, Itabashi-ku
  - Research Site, Shinjuku-ku

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ECU-MG-303&attachmentIdentifier=a5a00cf1-838d-459f-8838-a08248565a5f&fileName=ecu-mg-303-CSR_Synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included a Primary Evaluation Treatment Period of 26 weeks, an Extension Period of up to an additional 208 weeks, and a Follow-up Period of 8 weeks.
Pre-assignment Details: All participants were offered participation in the Extension Period of the study.
Groups:
- Eculizumab: Participants received eculizumab by intravenous (IV) infusion during the Primary Evaluation Treatment Period (26 weeks) and the Extension Period (up to 208 weeks). Dosing was initiated with a weekly weight-based induction regimen (Induction Phase) and, thereafter, participants were dosed every 2 weeks (Maintenance Phase). Eculizumab was administered at doses of 300, 600, 900, or 1200 milligrams (mg), based on the participant's current body weight.
Period: Primary Evaluation Period (26 Weeks)
Arm/Group | Eculizumab
Started | 11
Received at Least 1 Dose of Study Drug | 11 (Full Analysis Set/Safety Analysis Set)
Completed | 10
Not Completed | 1
Not completed — Physician Decision | 1
Period: Extension Period (Up to 208 Weeks)
Arm/Group | Eculizumab
Started | 10
Received at Least 1 Dose of Study Drug | 10 (Full Analysis Set)
Completed | 2
Not Completed | 8
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 1
Not completed — Participant transitioned to Ultomiris | 2
Not completed — Participant transitioned to Soliris | 1
Not completed — Participant transferred to another study | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who received at least 1 dose of eculizumab.
Groups:
- Eculizumab: Participants received eculizumab by IV infusion during the Primary Evaluation Treatment Period (26 weeks) and the Extension Period (up to 208 weeks). Dosing was initiated with a weekly weight-based induction regimen (Induction Phase) and, thereafter, participants were dosed every 2 weeks (Maintenance Phase). Eculizumab was administered at doses of 300, 600, 900, or 1200 mg, based on the participant's current body weight.
Arm/Group | Eculizumab
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.8 (1.78) [lower limit 1.78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1
Quantitative Myasthenia Gravis (QMG) Total Score [Mean (Standard Deviation); unit: units on a scale] — The QMG scoring system consists of 13 items: ocular (2 items), facial (1 item), bulbar (2 items), gross motor (6 items), axial (1 item), and respiratory (1 item). Each item is graded from 0 to 3, (0 = none, 1 = mild, 2 = moderate, and 3 = severe). The range of total QMG score is 0 to 39, with higher score indicating most severe disease.
  units on a scale | 16.7 (5.64) [lower limit 5.64]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the QMG Total Score at Week 26 Regardless of Rescue Treatment
Description: The QMG scoring system consists of 13 items: ocular (2 items), facial (1 item), bulbar (2 items), gross motor (6 items), axial (1 item), and respiratory (1 item). Each item is graded from 0 to 3, (0 = none, 1 = mild, 2 = moderate, and 3 = severe). The range of total QMG score is 0 to 39, with higher scores indicating more severe disease.
Time Frame: Baseline, Week 26
Population: Modified Full Analysis Set: all participants 12 to <18 years of age who received at least 1 dose of eculizumab. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eculizumab
Number analyzed (Participants) | 10
units on a scale | -6.1 (4.56) [lower limit 4.56]
Statistical Analysis 1: Comparison: Eculizumab; The observed change in QMG was analyzed with baseline QMG score and visits as covariates; Test type: Superiority; p = 0.0004, Repeated Measures Model; Least Square Mean = -5.8, 95% CI 2-sided [-8.40 to -3.13] — The least square mean change from baseline in QMG total score at Week 26 was calculated

2. Secondary Outcome: Change From Baseline in the Myasthenia Gravis Activities of Daily Living (MG-ADL) Total Score at Week 26 Regardless of Rescue Treatment
Description: The MG-ADL is an 8-point questionnaire that focuses on relevant symptoms and functional performance of activities of daily living in participants with myasthenia gravis (MG). The 8 items of the MG-ADL are derived from symptom-based components of the original 13-item QMG to assess disability secondary to ocular (2 items), bulbar (3 items), respiratory (1 item), and gross motor or limb (2 items) impairment related to effects from MG. In this functional status instrument, each response is graded from 0 (normal) to 3 (most severe). The range of total MG-ADL score is 0 to 24, with higher scores indicating more severe disease.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eculizumab
Number analyzed (Participants) | 10
units on a scale | -2.5 (1.78) [lower limit 1.78]

3. Secondary Outcome: Percentage of Participants With ≥3-Point Reduction in the MG-ADL Total Score With No Rescue Treatment
Description: The MG-ADL is an 8-point questionnaire that focuses on relevant symptoms and functional performance of activities of daily living in participants with MG. The 8 items of the MG-ADL are derived from symptom-based components of the original 13-item QMG to assess disability secondary to ocular (2 items), bulbar (3 items), respiratory (1 item), and gross motor or limb (2 items) impairment related to effects from MG. In this functional status instrument, each response is graded from 0 (normal) to 3 (most severe). The range of total MG-ADL score is 0 to 24, with higher scores indicating more severe disease.
Time Frame: Week 26
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 10
percentage of participants | 50.0 (18.7) [18.7 to 81.3]

4. Secondary Outcome: Percentage of Participants With ≥3-Point Reduction in the MG-ADL Total Score Regardless of Rescue Treatment
Description: as for outcome 3
Time Frame: Week 26
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 10
percentage of participants | 50.0 (18.7) [18.7 to 81.3]

5. Secondary Outcome: Percentage of Participants With ≥5-Point Reduction in the QMG Total Score With No Rescue Treatment
Description: as for outcome 1
Time Frame: Week 26
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 10
percentage of participants | 70.0 (34.8) [34.8 to 93.3]

6. Secondary Outcome: Percentage of Participants With ≥5-Point Reduction in the QMG Total Score Regardless of Rescue Treatment
Description: as for outcome 1
Time Frame: Week 26
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 10
percentage of participants | 70.0 (34.8) [34.8 to 93.3]

7. Secondary Outcome: Change From Baseline in the Myasthenia Gravis Composite (MGC) Scale Total Score at Week 26 Regardless of Rescue Treatment
Description: The MGC is a validated assessment tool for measuring clinical status of participants with MG. The MGC assesses 10 important functional areas most frequently affected by MG: ocular (2 items), facial (1 item), bulbar (3 items), respiratory (1 item), axial (1 item), and gross motor (2 items). The scales are weighted for clinical significance that incorporates patient-reported outcomes. The MGC total score ranges from 0 to 50, with lower scores indicating less functional impairment and higher scores indicating greater functional impairment.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eculizumab
Number analyzed (Participants) | 10
units on a scale | -9.4 (5.91) [lower limit 5.91]

8. Secondary Outcome: Change From Baseline in the European Quality of Life 5-Dimension Youth Version (EQ-5D-Y) Visual Analogue Scale (VAS) Score at Week 26 Regardless of Rescue Treatment
Description: The EQ-5D-Y is a reliable and validated survey of health status in 5 areas: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each of which is completed by the participant for participants ≥12 years of age (at time of assessment) and completed by the participant's caregiver or with caregiver assistance for participant <12 years of age. Each area has 3 levels: Level 1 (no problems), Level 2 (some problems), and Level 3 (extreme problems). The EQ visual analogue scale (VAS) records the participant's self-rated health on a vertical, 20-centimeter VAS where the endpoints are labelled 'Best imaginable health state, marked as 100' and 'Worst imaginable health state, marked as 0'.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eculizumab
Number analyzed (Participants) | 10
units on a scale | 23.5 (23.34) [lower limit 23.34]

9. Secondary Outcome: Change From Baseline in the Neurological Quality of Life-Fatigue Questionnaire (Neuro-QoL Pediatric Fatigue) Total Score at Week 26 Regardless of Rescue Treatment
Description: The Neuro-QoL Pediatric Fatigue questionnaire is a reliable and validated brief 11-item survey of fatigue, completed by the participant for participants ≥12 years of age (at time of assessment) and completed by the participant's caregiver or with caregiver assistance for participants <12 years of age. Each item was scored on a scale of 1 to 5 (1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=Very much). Total score is the sum of each item's score and it ranges from 11 to 55. Higher scores indicate greater fatigue and greater impact of MG on activities.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eculizumab
Number analyzed (Participants) | 10
units on a scale | -7.9 (7.37) [lower limit 7.37]

10. Secondary Outcome: Number of Participants in Each Category of the Myasthenia Gravis Foundation of America Post-Intervention Status (MGFAPIS) Regardless of Rescue Treatment at Week 26
Description: The MG clinical state (improved, unchanged, and worse) was assessed using the MGFAPIS.
Time Frame: Week 26
Population: Modified Full Analysis Set: all participants 12 to <18 years of age who received at least 1 dose of eculizumab. Here, 'Number Analyzed' and 'Overall Number of Participants Analyzed' signify those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 10
Participants
  Improved | 10
  Unchanged | 0
  Worse | 0

11. Secondary Outcome: Percentage of Participants With Clinical Deteriorations, Myasthenic Crises, and Rescue Therapy Use
Description: Rescue therapy (for example, high dose corticosteroid, plasma exchange, or intravenous immunoglobulin) was to be allowed when a participant experienced clinical deterioration. Clinical deterioration was defined as follows: Participants who experienced an MG crisis, which was defined as weakness due to MG that was severe enough to necessitate intubation or to delay extubation following surgery; or, Significant symptomatic worsening that required rescue medication in the opinion of the Investigator; or, Participants for whom the Investigator believed that the participants' health was in jeopardy if rescue therapy was not given.
Time Frame: Baseline up to Week 26
Population: Modified Full Analysis Set: all participants 12 to <18 years of age who received at least 1 dose of eculizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 11
percentage of participants
  Clinical Deterioration | 9.1
  MG Crisis | 9.1
  Requiring Rescue Therapy | 9.1

12. Secondary Outcome: Pharmacokinetics (PK): Serum Concentration Of Eculizumab
Time Frame: 24 hours postdose on Day 1; predose and 60 minutes postdose at Week 12; predose at Week 26
Population: Pharmacokinetic Analysis Set: all participants 12 to <18 years of age who received at least 1 dose of eculizumab and who had PK data assessments during the study. Here, 'Number Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms (μg)/milliliter (mL)
Arm/Group | Eculizumab
Number analyzed (Participants) | 11
micrograms (μg)/milliliter (mL)
  Day 1, 24 hours postdose | 359.6 (105.18)
  Week 12, Predose: number analyzed (Participants) | 10
  Week 12, Predose | 382.8 (159.57)
  Week 12, 60 minutes postdose | 910.5 (277.29)
  Week 26, Predose: number analyzed (Participants) | 9
  Week 26, Predose | 433.9 (171.85)

13. Secondary Outcome: Pharmacodynamics (PD): Serum Free Complement Component 5 Concentrations
Time Frame: Baseline; 24 hours postdose on Day 1; predose and 60 minutes postdose at Week 12; predose at Week 26
Population: Pharmacodynamic Analysis Set: all participants 12 to <18 years of age who received at least 1 dose of eculizumab and who had PD data assessments during the study. Here, 'Number Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Eculizumab
Number analyzed (Participants) | 11
μg/mL
  Baseline | 172.7 (34.52)
  Day 1, 24 hours postdose | 0.0 (0.01)
  Week 12, Predose | 0.0 (0.01)
  Week 12, 60 minutes postdose | 0.0 (0.01)
  Week 26, Predose: number analyzed (Participants) | 10
  Week 26, Predose | 0.0 (0.02)

14. Secondary Outcome: PD: Percentage of Hemolysis (In Vitro Assay)
Time Frame: Baseline; 24 hours postdose on Day 1; predose and 60 minutes postdose at Week 12; predose at Week 26
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage of hemolysis
Arm/Group | Eculizumab
Number analyzed (Participants) | 10
percentage of hemolysis
  Baseline | 105.8 (14.15)
  Day 1, 24 hours postdose | 1.1 (2.01)
  Week 12, Predose | 1.8 (4.67)
  Week 12, 60 minutes postdose | 0.2 (0.45)
  Week 26, Predose: number analyzed (Participants) | 9
  Week 26, Predose | 0.5 (1.29)

15. Secondary Outcome: Change From Baseline in the QMG Total Score at Week 52 Regardless of Rescue Treatment
Description: as for outcome 1
Time Frame: Baseline, Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eculizumab
Number analyzed (Participants) | 8
units on a scale | -4.9 (4.26) [lower limit 4.26]
Statistical Analysis 1: Comparison: Eculizumab; The observed change in QMG was analyzed with baseline QMG score and visits as covariates; Test type: Superiority; p = 0.0033, Repeated Measures Model; Least Square Mean = -4.3, 95% CI 2-sided [-6.93 to -1.65] — The least square mean change from baseline in QMG total score at Week 52 was calculated

ADVERSE EVENTS:
Time Frame: From date of first dose (Day 1) through 8 weeks after last dose (4 years and 7 months).
Description: Safety analysis set included all participants who received at least 1 dose of eculizumab.
Arm/Group | Eculizumab
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 4/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eculizumab (N=11)
Pyrexia (General disorders) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (8)
Myasthenia gravis crisis (Nervous system disorders) | 1 (2)
Suicide attempt (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Eculizumab (N=11)
Fatigue (General disorders) | 3 (5)
Infusion site extravasation (General disorders) | 1 (2)
Injection site bruising (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Vaccination site pain (General disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (10)
Upper respiratory tract infection (Infections and infestations) | 3 (4)
COVID-19 (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3)
Flatulence (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (21)
Nausea (Gastrointestinal disorders) | 1 (4)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 4 (16)
Dizziness (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Ketosis (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 2 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (1)
Monocytosis (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Glucose urine present (Investigations) | 1 (1)
Electrocardiogram PR prolongation (Investigations) | 1 (1)
Behaviour disorder (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (3)
Eye pruritus (Eye disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (2)
Ocular hyperaemia (Eye disorders) | 1 (1)
Device malfunction (Product Issues) | 1 (1)
Hypercalciuria (Renal and urinary disorders) | 1 (1)
Poor venous access (Vascular disorders) | 1 (1)
Pyrexia (General disorders) | 3 (8)
Immunisation reaction (Injury, poisoning and procedural complications) | 2 (2)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chronic fatigue syndrome (General disorders) | 1 (1)
Gait disturbances (General disorders) | 1 (1)
Infusion site discharge (General disorders) | 1 (1)
Infusion site swelling (General disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bicarbonate decreased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (1)
Post-traumatic headache (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asteatosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/9 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT03759366/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT03759366/SAP_002.pdf